CLINICAL TRIAL: NCT04575168
Title: Assess the Performance of Spartan COVID-19 V2 System in a Clinical Setting in Comparison to a Laboratory (Standard of Care (SOC)) PCR Method
Brief Title: Clinical Study Spartan COVID-19 V2 System
Status: Completed | Type: Observational
Sponsor: Spartan Bioscience Inc. (Industry)
Collaborators: Beaufort (Unknown)
Responsible Party: Sponsor
Other Study IDs: VNV-00615
Record Dates: First submitted 2020-10-01; First posted 2020-10-05 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive for COVID-19: Subjects positive for COVID-19 as indicated by the Standard of Care test.
  Interventions: Diagnostic Test: Spartan COVID-19 Test
- Negative for COVID-19: Subjects negative for COVID-19 as indicated by the Standard of Care test.
  Interventions: Diagnostic Test: Spartan COVID-19 Test

INTERVENTIONS:
Diagnostic Test: Spartan COVID-19 Test — A nasopharyngeal sample analyzed on the Spartan COVID-19 System.

SUMMARY:
This multicentre prospective study will enroll a sufficient number of patients to afford approximately 60 positives and > 40 negatives (as determined by the SOC - Comparator method) in the United States and/or Canada. One to three sites in the United States and/or Canada will participate over an approximate 12-week enrolment period. The actual enrolment period will be dependent upon prevalence of Covid-19. Once positives sample size is achieved, expected SARC-CoV-2 negative subjects will be permitted.

This study is observational and will not impact the medical management of the patient. The results of the Spartan Test will be blinded to the clinical staff during the study and will not impact the medical management of the subject.

Once informed consent is obtained and eligibility is confirmed, subject demographics, and patient reported COVID-19 symptoms will be recorded. For the purposes of this study, enrolment will be defined as the collection of the two study-specific nasopharyngeal (NP) samples for Spartan's Test. Each patient's active involvement in the study will last for approximately 30 minutes.

To support the EUA, a minimum of 30 individual natural positive clinical specimens will be collected from patients suspected of SARS-CoV-2 infection by a healthcare provider in COVID-19 disease endemic regions in the United States. Additionally, a minimum of 30 individual negative samples will also be used to support the EUA from patients in the United States.

Once subjects are consented and recruited for the study, three nasopharyngeal samples for each patient will be collected by trained operators at the clinical site. The first sample will be tested at the clinical site according to standard of care protocols currently in place for the sites' nasopharyngeal swab-based SARS-CoV-2 RT-PCR testing. The second nasopharyngeal sample will be tested at the site using the Spartan COVID-19 v2 System. The third nasopharyngeal sample will be tested using the Spartan COVID-19 v2 System only when the test conducted with the second nasopharyngeal swab does not produce a positive or negative result.

The sample for the SOC test will be collected prior to the samples for the Spartan COVID-19 v2 System as per clinical regulations.

ELIGIBILITY:
Inclusion Criteria:

* Individuals suspected of SARS-CoV-2 infection by a healthcare provider
* Individuals whose first symptom onset occurred less than or equal to 7 days of presentation
* Individual (or authorized representative) able or willing to provide written informed consent for study participation

Exclusion Criteria:

* Vulnerable populations (e.g., women with pregnancy, institutionalized individual) as deemed inappropriate for study by the site investigator
* Individuals with self-reported nosebleed within 24 hours of presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting to clinical study sites with symptoms of SARS-CoV-2 or suspected of SARS-Cov-2 infection by a healthcare provider
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Percent Agreement between SOC test and Spartan COVID-19 test | 24hours
  Overall percent agreement between the test results generated by the Spartan COVID-19 v2 System and the nasopharyngeal swab-based SARS-Cov-2 test currently in use at the clinical site (SOC test)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Wake Research Mt. Vernon, Sandy Springs, Georgia
  - Clinical Chemistry Research Lab, University of Maryand-Baltimore, Baltimore, Maryland
  - Wake Research ClinSearch, Chattanooga, Tennessee